CLINICAL TRIAL: NCT04679805
Title: Impact of Coronary Angioplasty on Non-hyperaemic Pressure Ratio in Patients With Coronary Artery Disease.
Brief Title: Physio PCI: Impact of Coronary Angioplasty on Non-hyperaemic Pressure Ratio in Patients With Coronary Artery Disease
Status: Terminated | Type: Observational
Why Stopped: Due to COVID-19 pandemic site refused to include patients in the study
Sponsor: Ceric Sàrl (Industry)
Responsible Party: Sponsor
Other Study IDs: Physio PCI Study
Record Dates: First submitted 2020-12-17; First posted 2020-12-22 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Coronary Artery Disease
Keywords: Percutaneous Coronary Intervention; Fractional Flow Reserve; Resting Full Cycle Ratio
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The use of intra coronary physiological assessment with fractional flow reserve (FFR) is nowadays the standard approach to define ischemia-inducing stenosis and guide myocardial revascularization strategy in patients with coronary artery disease. Further, FFR has been shown to be a strong and independent predictor of major adverse cardiac events after stent implantation. A lower value of FFR after stent implantation is associated with a worse clinical prognosis, without a clearly defined threshold above which clinical follow up are similar for all FFR values. Among 750 patients in the Fractional Flow Reserve Post-Stent Registry, the event rate was 29.5% in patients with FFR<0.80 compared to 9 4.9% in patients with FFR>0.95 (p<0.001). However, FFR remains poorly adopted in many cathlabs, partly because of procedural time, discomfort or sides effect during hyperemia, non-uniform adenosine response and economical constraints. This leads to the validation of resting indices (instantaneous wave-free ratio (iFR), diastolic pressure ratio (dPR), and resting full-cycle ratio (RFR) among others). Those indices evaluate coronary physiology without the use of maximal hyperemia and have 15 slightly different threshold compared to FFR (≤0.89 vs 0.80, for iFR and RFR, and FFR 16 respectively).In the VALIDATE RFR study, a head-to-head comparison of RFR and iFR from a retrospective analysis, diagnostic accuracy of RFR was 97.4% with an area under the curve 1 (AUC) of 99.6%. In the more recent RE-VALIDATE RFR study, 431 patients with 501 lesions 2 were prospectively evaluated for the diagnostic performance of RFR in all-comers patients. Compared to iFR, RFR achieved high diagnostic accuracy, sensitivity and specificity. These are the reasons why we designed a prospective, non-randomized, clinical trial, to better 18 explore the value of RFR before and after PCI in real live and after optimization by post dilation 19 in all-comers patients with coronary artery disease in the Middle East region..

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 21 years
* The patient is deemed eligible for PCI of at least one coronary stenosis (RFRpre ≤0.89 or FFR≤0.80)
* The patient is able and is willing to comply with all study procedures and process.

Exclusion Criteria:

* The patient is in cardiogenic shock
* The patient has a bifurcation lesion that requires a planned two stents technique
* The patient refuses to participate.
* The patient suffers acute coronary syndrome and should be treated by PCI in the culprit lesion (non-culprit lesions in non-culprit vessel could be included)
* The patient has an ostial stenosis to be treated by PCI

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female subjects could be enrolled in the present study if they are 21 years old or older at the time of inclusion. The trial will enroll 100 patients who need to meet ALL eligibility criteria and provide written informed consent prior to inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2021-06-06 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
RFRpre vs. RFRfinal | Intra operative, up to 1 month
  comparison between RFR (Resting Full Cycle Ratio) before and after optimized PCI (RFRpre vs. RFRfinal) in all included lesions

SECONDARY OUTCOMES:
RFRpre vs. RFRpost | Intra operative, up to 1 month
  Comparison of RFR (Resting Full Cycle Ratio) value before and after PCI
RFRpost vs. RFRfinal | Intra operative, up to 1 month
  Comparison of RFR (Resting Full Cycle Ratio) value before and after PCI optimization
FFRpre vs. FFRpost | Intra operative, up to 1 month
  Comparison of FFR (Fractional Flow reserve) value before and after PCI
FFRpost vs. FFRfinal | Intra operative, up to 1 month
  Comparison of FFR (Fractional Flow reserve) value before and after optimized PCI
FFRpre vs. FFRfinal | Intra operative, up to 1 month
  Comparison of FFR (Fractional Flow reserve) value before and after PCI
RFRpre vs. FFRpre: % of lesions | Intra operative, up to 1 month
  Comparison of FFR (Fractional Flow reserve) and RFR (Resting Full Cycle Ratio) value before PCI: % of lesions with FFR≤0.80 compared to RFR≤0.89.
RFRpost vs. FFRpost/ % of lesions | Intra operative, up to 1 month
  Comparison of FFR (Fractional Flow reserve) and RFR (Resting Full Cycle Ratio) value after PCI : % of lesions with FFR≤0.80 compared to RFR≤0.89
RFRfinal vs. FFRfinal/ % of lesions | Intra operative, up to 1 month
  Comparison of FFR (Fractional Flow reserve) and RFR (Resting Full Cycle Ratio) value after optimized PCI : % of lesions with FFR≤0.80 compared to RFR≤0.89.
Proc Timepost vs. Proc Timefinal. | Intra operative, up to 1 month
  Duration of the procedure (mn) after PCI optimization
Irradiationpost vs. Irradiationfinal. | Intra operative, up to 1 month
  Irradiation during the procedure in mGy after PCI and after optimization:
Contrastpost vs. Contrastfinal. | Intra operative, up to 1 month
  Volume of contrast dye load (cc) during the procedure after PCI and after optimization
% of patients: RFRpost vs. RFRfinal | Intra operative, up to 1 month
  % of patients with (Resting Full Cycle Ratio) RFR > 0.70, 0.80, 0.89 and 0.95 (in the treated vessel in case of 1 multivessel CAD) before and after optimization
The rate of Major Adverse Coronary Events | Day 1 and Day 30
  Major Adverse Coronary Events: cardiovascular mortality, myocardial infarction, ischemia driven target lesion revascularization
The rate of all cause mortality | Day 1 and Day 30
  All-cause mortality
The rate of Stent Thrombosis | Day 1 and Day 30
  Stent thrombosis according to the definition of ARC2 (definite or probable)

CONTACTS AND LOCATIONS:
Overall Officials: Arif Al Nooryani, Principal Investigator — Al Qassimi Hospital
Locations (1):
- Al Qassimi Hospital, Sharjah city, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Neumann FJ, Sousa-Uva M, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO; ESC Scientific Document Group. 2018 ESC/EACTS Guidelines on myocardial revascularization. Eur Heart J. 2019 Jan 7;40(2):87-165. doi: 10.1093/eurheartj/ehy394. No abstract available. PMID 30165437
- [Result] Fearon WF, Luna J, Samady H, Powers ER, Feldman T, Dib N, Tuzcu EM, Cleman MW, Chou TM, Cohen DJ, Ragosta M, Takagi A, Jeremias A, Fitzgerald PJ, Yeung AC, Kern MJ, Yock PG. Fractional flow reserve compared with intravascular ultrasound guidance for optimizing stent deployment. Circulation. 2001 Oct 16;104(16):1917-22. doi: 10.1161/hc4101.097539. PMID 11602494
- [Result] Pijls NH, Klauss V, Siebert U, Powers E, Takazawa K, Fearon WF, Escaned J, Tsurumi Y, Akasaka T, Samady H, De Bruyne B; Fractional Flow Reserve (FFR) Post-Stent Registry Investigators. Coronary pressure measurement after stenting predicts adverse events at follow-up: a multicenter registry. Circulation. 2002 Jun 25;105(25):2950-4. doi: 10.1161/01.cir.0000020547.92091.76. PMID 12081986
- [Result] Doh JH, Nam CW, Koo BK, Lee SY, Choi H, Namgung J, Kwon SU, Kwak JJ, Kim HY, Choi WH, Lee WR. Clinical Relevance of Poststent Fractional Flow Reserve After Drug-Eluting Stent Implantation. J Invasive Cardiol. 2015 Aug;27(8):346-51. PMID 26232010
- [Result] Agarwal SK, Kasula S, Hacioglu Y, Ahmed Z, Uretsky BF, Hakeem A. Utilizing Post-Intervention Fractional Flow Reserve to Optimize Acute Results and the Relationship to Long-Term Outcomes. JACC Cardiovasc Interv. 2016 May 23;9(10):1022-31. doi: 10.1016/j.jcin.2016.01.046. PMID 27198682
- [Result] Li SJ, Ge Z, Kan J, Zhang JJ, Ye F, Kwan TW, Santoso T, Yang S, Sheiban I, Qian XS, Tian NL, Rab TS, Tao L, Chen SL. Cutoff Value and Long-Term Prediction of Clinical Events by FFR Measured Immediately After Implantation of a Drug-Eluting Stent in Patients With Coronary Artery Disease: 1- to 3-Year Results From the DKCRUSH VII Registry Study. JACC Cardiovasc Interv. 2017 May 22;10(10):986-995. doi: 10.1016/j.jcin.2017.02.012. Epub 2017 Apr 26. PMID 28456699
- [Result] Hwang D, Lee JM, Lee HJ, Kim SH, Nam CW, Hahn JY, Shin ES, Matsuo A, Tanaka N, Matsuo H, Lee SY, Doh JH, Koo BK. Influence of target vessel on prognostic relevance of fractional flow reserve after coronary stenting. EuroIntervention. 2019 Aug 29;15(5):457-464. doi: 10.4244/EIJ-D-18-00913. PMID 30561367
- [Result] Davies JE, Sen S, Dehbi HM, Al-Lamee R, Petraco R, Nijjer SS, Bhindi R, Lehman SJ, Walters D, Sapontis J, Janssens L, Vrints CJ, Khashaba A, Laine M, Van Belle E, Krackhardt F, Bojara W, Going O, Harle T, Indolfi C, Niccoli G, Ribichini F, Tanaka N, Yokoi H, Takashima H, Kikuta Y, Erglis A, Vinhas H, Canas Silva P, Baptista SB, Alghamdi A, Hellig F, Koo BK, Nam CW, Shin ES, Doh JH, Brugaletta S, Alegria-Barrero E, Meuwissen M, Piek JJ, van Royen N, Sezer M, Di Mario C, Gerber RT, Malik IS, Sharp ASP, Talwar S, Tang K, Samady H, Altman J, Seto AH, Singh J, Jeremias A, Matsuo H, Kharbanda RK, Patel MR, Serruys P, Escaned J. Use of the Instantaneous Wave-free Ratio or Fractional Flow Reserve in PCI. N Engl J Med. 2017 May 11;376(19):1824-1834. doi: 10.1056/NEJMoa1700445. Epub 2017 Mar 18. PMID 28317458
- [Result] Gotberg M, Christiansen EH, Gudmundsdottir IJ, Sandhall L, Danielewicz M, Jakobsen L, Olsson SE, Ohagen P, Olsson H, Omerovic E, Calais F, Lindroos P, Maeng M, Todt T, Venetsanos D, James SK, Karegren A, Nilsson M, Carlsson J, Hauer D, Jensen J, Karlsson AC, Panayi G, Erlinge D, Frobert O; iFR-SWEDEHEART Investigators. Instantaneous Wave-free Ratio versus Fractional Flow Reserve to Guide PCI. N Engl J Med. 2017 May 11;376(19):1813-1823. doi: 10.1056/NEJMoa1616540. Epub 2017 Mar 18. PMID 28317438
- [Result] Svanerud J, Ahn JM, Jeremias A, van 't Veer M, Gore A, Maehara A, Crowley A, Pijls NHJ, De Bruyne B, Johnson NP, Hennigan B, Watkins S, Berry C, Oldroyd KG, Park SJ, Ali ZA. Validation of a novel non-hyperaemic index of coronary artery stenosis severity: the Resting Full-cycle Ratio (VALIDATE RFR) study. EuroIntervention. 2018 Sep 20;14(7):806-814. doi: 10.4244/EIJ-D-18-00342. PMID 29790478
- [Result] Lee JM, Choi KH, Park J, Hwang D, Rhee TM, Kim J, Park J, Kim HY, Jung HW, Cho YK, Yoon HJ, Song YB, Hahn JY, Nam CW, Shin ES, Doh JH, Hur SH, Koo BK. Physiological and Clinical Assessment of Resting Physiological Indexes. Circulation. 2019 Feb 12;139(7):889-900. doi: 10.1161/CIRCULATIONAHA.118.037021. PMID 30586749
- [Result] Mallidi J, Atreya AR, Cook J, Garb J, Jeremias A, Klein LW, Lotfi A. Long-term outcomes following fractional flow reserve-guided treatment of angiographically ambiguous left main coronary artery disease: A meta-analysis of prospective cohort studies. Catheter Cardiovasc Interv. 2015 Jul;86(1):12-8. doi: 10.1002/ccd.25894. Epub 2015 Mar 19. PMID 25676445
- [Result] Shaheen M, Mokarrab M, Youssef A, Aref M, Abushouk AI, Elmaraezy A, Almasswary A. Physiological evaluation of the provisional side-branch intervention strategy for bifurcation lesions using instantaneous wave-free ratio. Indian Heart J. 2018 Dec;70 Suppl 3(Suppl 3):S254-S258. doi: 10.1016/j.ihj.2018.01.028. Epub 2018 Jan 31. PMID 30595269
- [Result] Kobayashi Y, Johnson NP, Berry C, De Bruyne B, Gould KL, Jeremias A, Oldroyd KG, Pijls NHJ, Fearon WF; CONTRAST Study Investigators. The Influence of Lesion Location on the Diagnostic Accuracy of Adenosine-Free Coronary Pressure Wire Measurements. JACC Cardiovasc Interv. 2016 Dec 12;9(23):2390-2399. doi: 10.1016/j.jcin.2016.08.041. Epub 2016 Nov 9. PMID 27838269
- [Result] van Zandvoort LJC, Masdjedi K, Witberg K, Ligthart J, Tovar Forero MN, Diletti R, Lemmert ME, Wilschut J, de Jaegere PPT, Boersma E, Zijlstra F, Van Mieghem NM, Daemen J. Explanation of Postprocedural Fractional Flow Reserve Below 0.85. Circ Cardiovasc Interv. 2019 Feb;12(2):e007030. doi: 10.1161/CIRCINTERVENTIONS.118.007030. PMID 30732469
- [Result] Meneveau N, Souteyrand G, Motreff P, Caussin C, Amabile N, Ohlmann P, Morel O, Lefrancois Y, Descotes-Genon V, Silvain J, Braik N, Chopard R, Chatot M, Ecarnot F, Tauzin H, Van Belle E, Belle L, Schiele F. Optical Coherence Tomography to Optimize Results of Percutaneous Coronary Intervention in Patients with Non-ST-Elevation Acute Coronary Syndrome: Results of the Multicenter, Randomized DOCTORS Study (Does Optical Coherence Tomography Optimize Results of Stenting). Circulation. 2016 Sep 27;134(13):906-17. doi: 10.1161/CIRCULATIONAHA.116.024393. Epub 2016 Aug 29. PMID 27573032
- [Result] Thygesen K, Alpert JS, Jaffe AS, Chaitman BR, Bax JJ, Morrow DA, White HD; Executive Group on behalf of the Joint European Society of Cardiology (ESC)/American College of Cardiology (ACC)/American Heart Association (AHA)/World Heart Federation (WHF) Task Force for the Universal Definition of Myocardial Infarction. Fourth Universal Definition of Myocardial Infarction (2018). J Am Coll Cardiol. 2018 Oct 30;72(18):2231-2264. doi: 10.1016/j.jacc.2018.08.1038. Epub 2018 Aug 25. No abstract available. PMID 30153967
- [Result] Cutlip DE, Windecker S, Mehran R, Boam A, Cohen DJ, van Es GA, Steg PG, Morel MA, Mauri L, Vranckx P, McFadden E, Lansky A, Hamon M, Krucoff MW, Serruys PW; Academic Research Consortium. Clinical end points in coronary stent trials: a case for standardized definitions. Circulation. 2007 May 1;115(17):2344-51. doi: 10.1161/CIRCULATIONAHA.106.685313. PMID 17470709